CLINICAL TRIAL: NCT05763628
Title: Performance Evaluation of Different Daily Disposable Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-144
Record Dates: First submitted 2023-02-21; First posted 2023-03-10 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-03

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens, then Test Lens (Experimental): Participants wore Control Lens for 2 weeks, then crossed over to Test Lens for 2 weeks.
  Interventions: Device: Control Lens (stenfilcon A); Device: Test Lens (senofilcon A)
- Test Lens, then Control Lens (Experimental): Participants wore Test Lens for 2 weeks, then crossed over to Control Lens for 2 weeks.
  Interventions: Device: Control Lens (stenfilcon A); Device: Test Lens (senofilcon A)

INTERVENTIONS:
Device: Control Lens (stenfilcon A) — Daily Disposable Multifocal Contact Lens for 2 weeks
Device: Test Lens (senofilcon A) — Daily Disposable Multifocal Contact Lens for 2 weeks

SUMMARY:
The objective of the study was to compare the lens performance of two daily disposable multifocal contact lenses.

DETAILED DESCRIPTION:
This was a prospective, randomized, participant-masked, crossover, bilateral dispensing study. Each lens type was worn for approximately 3-4 weeks: the lens prescription of each lens type was optimized after a 3-8 days wearing experience, then participants began a 2 week (14-21 day) wear period.

ELIGIBILITY:
Inclusion Criteria:

1. Were at least 42 years of age and had full legal capacity to volunteer;
2. Had read and signed an information consent letter;
3. Self-reported having had a full eye examination in the previous two years;
4. Anticipated being able to wear the study lenses for at least 8 hours a day, 5 days a week
5. Were willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wore multifocal soft contact lenses, for the past 3 months minimum

   * Maximum of 7 participants per site were habitual wearers of daily disposable lenses
   * Maximum of 3 habitual wearers per site of 1-Day Acuvue Moist Multifocal
   * Maximum of 1 habitual wearer per site of ACUVUE OASYS MAX 1-Day MULTIFOCAL
   * Maximum of 3 habitual wearers per site of MyDay Multifocal
   * Maximum of 7 participants per site were habitual wearers of frequent replacement lenses
   * Maximum of 1 habitual wearer per site of ACUVUE OASYS for PRESBYOPIA
7. Had refractive astigmatism no higher than -0.75DC in each eye;
8. Were presbyopic and required a reading addition of at least +0.75D and no more than +2.50D;
9. Could be fit and achieved binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deemed to be 'acceptable', with the available study lens parameters (powers +4.00 to -6.00DS, near addition as per study design)

Exclusion Criteria:

A person was excluded from the study if they:

1. Were participating in any concurrent clinical or research study;
2. Had any known active ocular disease and/or infection that contraindicated contact lens wear;
3. Had a systemic condition that in the opinion of the investigator may have affected a study outcome variable;
4. Were using any systemic or topical medications that in the opinion of the investigator may have affected contact lens wear or a study outcome variable;
5. Had known sensitivity to the diagnostic sodium fluorescein to be used in the study;
6. Self-reported as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Had undergone refractive error surgery or interocular surgery.

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wilkinson, Principal Investigator — Spadina Optometry; Ashley Tucker, Principal Investigator — Bellaire Family Eye Care; Fiona Soong, Principal Investigator — Eyes on Sheppard Clinic; Andrew Sacco, Principal Investigator — Sacco Eye Group PLLC; Shane Foster, Principal Investigator — Athens Eye Care - Dr. Shane Foster & Associates
Locations (5):
- United States (3):
  - Sacco Eye Group PLLC, Vestal, New York
  - Athens Eye Care- Dr. Shane Foster & Associates, Athens, Ohio
  - Bellaire Family Eye Care, Bellaire, Texas
- Canada (2):
  - Eyes on Sheppard Clinic, Toronto, Ontario
  - Spadina Optometry, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 60 participants screened, 1 exited the study prior to randomization due to screen failure.
Groups:
- Control Lens, Then Test Lens: Participants first wore Control Lens for 2 weeks, then crossed over to wear Test Lens for 2 weeks
- Test Lens, Then Control Lens: Participants first wore Test Lens for 2 weeks, then crossed over to wear Control Lens for 2 weeks
Period: Period 1: First Intervention, 2 Weeks
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 29 | 30
Completed | 29 | 28
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2: Second Intervention, 2 Weeks
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 29 | 28
Completed | 28 | 28
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were screened for the study. Baseline data was collected from participants not considered Enrolled in the study.
Groups:
- Total Study Population: All participants that attended one or more study visits
Arm/Group | Total Study Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling for Removal
Description: Subjective rating for ease of removal of the study lenses on a 0-100 scale, where 0=Very difficult and 100=Very easy. Collected once at the end of 2 weeks of wear.
Time Frame: 2 Weeks
Population: Participants that completed all study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Lens: Participants that received the Control Lens during either the first or second period of the study
- Test Lens: Participants that received the Test Lens during either the first or second period of the study
Arm/Group | Control Lens | Test Lens
Number analyzed (Participants) | 56 | 56
score on a scale | 94 (10) | 95 (10)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 6 weeks (prescription optimization for 3-8 days, then test lens wear for 2 weeks each)
Arm/Group | Control Lens | Test Lens
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/58
Other Adverse Events (participants affected / at risk) | 2/57 | 3/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Lens (N=57) | Test Lens (N=58)
Stye (Eye disorders) | 0 (0) | 1 (1)
Eyelid myokymia (Eye disorders) | 1 (1) | 0 (0)
Dose increase (Surgical and medical procedures) | 0 (0) | 1 (1) — Urologist increased dosage of current medication. Non-ocular and unrelated to study lens.
Botox Injection Forehead (Surgical and medical procedures) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT05763628/Prot_SAP_000.pdf